CLINICAL TRIAL: NCT07092735
Title: Optimizing Elite Football Performance Through Neuro-Athletic Training: A Parallel-Group Randomized Controlled Trial
Brief Title: Neuro-Athletic Training in Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/71
Record Dates: First submitted 2025-07-09; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Athletic Performance; Neurocognitive Function; Proprioception; Soccer; Sensorimotor Integration; Eye Movements; Neuroathletic Training

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group randomized controlled trial design with pre- and post-intervention assessments. Participants were randomly assigned to either a Neuro-Athletic Training (NAT) group or a control group. The NAT group received an 8-week structured program targeting sensorimotor integration through oculomotor, vestibular, and proprioceptive drills, while the control group continued standard football training without additional interventions. Outcome assessors and statistical analysts were blinded to group allocations. The study was conducted under standardized conditions to ensure methodological rigor and group comparability.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments were performed by an independent physiotherapist who was blinded to group allocation to reduce measurement bias. Additionally, the researcher conducting the statistical analysis was also blinded to group assignments to ensure data objectivity. Participants and intervention providers were not blinded due to the nature of the behavioral intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-Athletic Training (NAT) Group (Experimental): Participants receive a structured 8-week NAT program including oculomotor, vestibular, and proprioceptive drills, 3 sessions/week (35-45 minutes each).
  Interventions: Behavioral: Neuro-Athletic Training
- Standard Training Group (Active Comparator): Participants continue their standard in-season football training program without any NAT components.
  Interventions: Other: Standard Training

INTERVENTIONS:
Behavioral: Neuro-Athletic Training — Participants receive a structured 8-week NAT program including oculomotor, vestibular, and proprioceptive drills, 3 sessions/week (35-45 minutes each).
  Arms: Neuro-Athletic Training (NAT) Group
Other: Standard Training — Participants continue their standard in-season football training program without any NAT components.
  Arms: Standard Training Group

SUMMARY:
This randomized controlled trial evaluates the effectiveness of an 8-week neuro-athletic training (NAT) program in enhancing sport-specific skills and physical capacities in elite male football players aged 18-23 years. Participants were randomly assigned to a NAT intervention group or a control group that maintained standard training. The NAT program involved oculomotor, vestibular, and proprioceptive drills. Primary outcomes include passing and shooting accuracy; secondary outcomes include flexibility and isokinetic knee strength.

ELIGIBILITY:
Inclusion Criteria:

* Male football players aged 18-23 years
* Active in the Turkish Regional Amateur League (2023-2024 season)
* Minimum of 5 years of uninterrupted football training experience
* No known neuromuscular or visual impairments
* Participation in at least four football training sessions per week
* Willingness and ability to participate in all assessments and training sessions
* Provision of written informed consent

Exclusion Criteria:

* History of orthopedic or neurological surgery within the past year
* Acute or chronic musculoskeletal injuries preventing full participation
* Uncorrected visual impairment
* Use of medications affecting neuromuscular performance or coordination
* Previous or concurrent involvement in structured neuromuscular or neuro-athletic training programs
* Irregular attendance to training sessions (>20% missed)
* Any condition precluding safe participation, as determined by medical staff

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as male are eligible to participate in this study. The study targets elite male football players to ensure homogeneity in performance characteristics and to align with league-specific demographics during the 2023-2024 season.
Enrollment: 56 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Passing Accuracy (Mor-Christian Passing Test) | Pre-intervention (baseline) and post-intervention (after 8 weeks).
  Measured as a score (max 120) based on 12 passes from 7, 8.5, and 10 meters toward a mini-goal. Assessed pre- and post-intervention.
Shooting Accuracy (Mor-Christian Shooting Test) | Pre-intervention (baseline) and post-intervention (after 8 weeks).
  Measured as a score (max 80) based on 16 shots from 14.5 meters toward four 45 cm targets. Assessed pre- and post-intervention.

SECONDARY OUTCOMES:
Flexibility (Sit-and-Reach Test) | Pre-intervention (baseline) and post-intervention (after 8 weeks)
  Measured in centimeters using a standard sit-and-reach box, assessing hamstring and lower back flexibility.
Isokinetic Knee Strength (ISOMED 2000 Dynamometer) | Pre-intervention (baseline) and post-intervention (after 8 weeks).
  Concentric peak torque of quadriceps and hamstrings at 60°/s (5 repetitions) and 180°/s (15 repetitions), normalized to body mass (Nm/kg), and hamstring-to-quadriceps (H:Q) ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional data protection policies.